CLINICAL TRIAL: NCT03276923
Title: Maternal Autoimmune Disease Research Alliance (MADRA) Registry
Acronym: MADRA
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00084014
Record Dates: First submitted 2017-08-29; First posted 2017-09-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Autoimmune Diseases; Pregnancy Related; Systemic Lupus Erythematosus; Cutaneous Lupus; Rheumatoid Arthritis; Sjogren's Syndrome; Scleroderma
MeSH Terms: conditions — Autoimmune Diseases; Lupus Erythematosus, Systemic; Arthritis, Rheumatoid; Sjogren's Syndrome; Scleroderma, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 100 Years
Biospecimen Retention: Samples With DNA — Blood and urine samples will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Maternal Autoimmune Disease ReseArch (MADRA) Registry: Women with autoimmune diseases who are pregnant

SUMMARY:
This multi-site registry, centered at Duke University, will enroll pregnant women with autoimmune and rheumatologic diseases.

The main goal of MADRA is to identify ways to improve the health of women with rheumatic diseases and their babies during pregnancy.

Prior studies demonstrate the importance of increase inflammation prior to and during pregnancy on these outcomes. The future research will seek to better define these risk factors and to identify ways to may improve them.

DETAILED DESCRIPTION:
At each site, the patients will be under the care of the participating rheumatologist and their local obstetrician during the pregnancy. This is a natural-history study and will not include medications, laboratory testing, or procedures outside of the standard of care.

Management of the rheumatologic disease will be directed based on patient needs by the local rheumatologist and obstetrician. Enrollment in the registry will not dictate specific therapy. The Registry will include data from each office visit during pregnancy and up to 12 months after delivery.

The registry will be ongoing, with periodic analysis of clinical data samples as specific studies are approved.

Enrollment in the registry does not significantly increase risks for a patient.

ELIGIBILITY:
Inclusion Criteria:

* Desire for pregnancy within 6 months or currently pregnant
* Women with systemic autoimmune disease, including:
* Lupus (systemic lupus erythematosus or cutaneous lupus)
* Antiphospholipid Syndrome or positive antiphospholipid antibodies
* Rheumatoid Arthritis
* Scleroderma (systemic sclerosis)
* Sjogren's Syndrome
* Inflammatory Arthritis (including Psoriatic Arthritis and Ankylosing Spondylitis)
* Undifferentiated Connective Tissue Disease (UCTD)
* Vasculitis
* Myositis (Polymyositis or Dermatomyositis)
* Positive Ro/SSA or La/SSB antibodies

Exclusion Criteria:

* Unable to speak English
* Unable to provide informed consent
* Unable to travel to Duke University for follow-up visits

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Women who have been diagnosed with an autoimmune disease or a rheumatic condition.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Risk factors associated with poor pregnancy outcomes as measured by the MADRA-DAP questionnaire. | up to 10 years
  The investigators will ask the participants questions from the MADRA-DAP questionnaire to determine poor pregnancy outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Megan EB Clowse, MD, MPH, Principal Investigator — Duke Health
Locations (1):
- Duke University, Durham, North Carolina, United States